CLINICAL TRIAL: NCT06191640
Title: Sinus Disease in Young Children With Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Kansas Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Iowa (Other); University of Virginia (Other); University of Vermont (Other); University of North Carolina, Chapel Hill (Other); Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Daniel M. Beswick, MD; Associate Professor-in-Residence; Associate Residency Program Director; Co-Chair, Equity, Diversity, and Inclusion Committee Department of Head and Neck Surgery, University of California, Los Angeles
Other Study IDs: 22-000594
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis in Children; Cystic Fibrosis; Chronic Rhinosinusitis (Diagnosis); Olfactory Disorder; Olfactory Impairment
Keywords: Cystic Fibrosis; Chronic Rhinosinusitis; Olfactory Dysfunction
MeSH Terms: conditions — Cystic Fibrosis; Disease; Olfaction Disorders | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HEMT Group: Children with CF planning to start ivacaftor or elexacaftor/tezacaftor/ivacaftor CFTR modulator therapy. Participants from the non-HEMT group of this study may enroll into the HEMT cohort if they become eligible for these CFTR modulator therapies and plan to start them.
  Interventions: Drug: Ivacaftor or elexacaftor/tezacaftor/ivacaftor
- Non-HEMT/Control Group: Children with CF not on ivacaftor or elexacaftor/tezacaftor/ivacaftor CFTR modulator therapy.

INTERVENTIONS:
Drug: Ivacaftor or elexacaftor/tezacaftor/ivacaftor — HEMT's are prescribed at the discretion of the treating physician and is not dictated by the principal investigator of this study.
  Other Names: Kalydeco or Trikafta; Vertex (VX)-770 or VX-445/VX-661/VX-770
  Groups: HEMT Group

SUMMARY:
This is a prospective, observational study examining the impact of highly effective cystic fibrosis transmembrane conductance regulator (CFTR) modulators on chronic rhinosinusitis (CRS) and olfactory dysfunction (OD) in young children with cystic fibrosis (YCwCF). This study involves two groups: children 2-8 years old, inclusive at initial visit, receiving highly effective modulator therapy (HEMT), and a control group of children 2-8 years old, inclusive at initial visit, not receiving HEMT. Outcomes will include sinus magnetic resonance imaging (MRI) scans, olfactory tests, and quality of life surveys obtained over a two-year period.

DETAILED DESCRIPTION:
This multi-center, prospective, observational study investigates the effects of highly effective modulator therapy (HEMT) on chronic rhinosinusitis (CRS) and olfactory dysfunction (OD) in young children with cystic fibrosis (YCwCF). The study spans two years and includes two distinct groups of children with cystic fibrosis: children ≤ 8 years old receiving HEMT and a control group of children ≤ 8 not receiving HEMT. The study aims to assess the efficacy of HEMT in improving sinus health and olfactory capabilities in this young demographic.

Key assessments include magnetic resonance imaging (MRI) sinus opacification, olfactory bulb volume measured via MRI, objective olfactory testing, and various quality (QOL) surveys. This investigation seeks to characterize the severity of CRS and OD in YCwCF, and to elucidate if early initiation of HEMT improves CRS and OD .

In the HEMT group, participants will have a pre-HEMT assessment followed by 1-year and 2-year post-HEMT evaluations. In the control/non-HEMT group, participants will undergo parallel assessments at baseline, 1-year, and 2-year intervals to track the natural progression of CRS and OD without HEMT.

ELIGIBILITY:
Inclusion Criteria:

HEMT Group:

* Children with documentation of a CF diagnosis
* Age 2-8 years old at first study visit
* CFTR mutation consistent with FDA labeled indication of highly effective modulator therapy (ivacaftor or elexacaftor/tezacaftor/ivacaftor)
* Clinician intent to prescribe ivacaftor or ETI so that enrollment is before start of HEMT

Non-HEMT/Control Group:

* Children with documentation of a CF diagnosis
* Age 2-8 years at first study visit
* Ineligible for highly effective modulator therapy (ivacaftor or elexacaftor/tezacaftor/ivacaftor) based on CFTR mutation or clinical decision not to initiate HEMT if eligible

Exclusion Criteria:

For Both Groups:

* Use of an investigational drug within 28 days prior to the first study visit
* Use of ivacaftor or elexacaftor/tezacaftor/ivacaftor within the 180 days prior to and including the first study visit
* Use of chronic oral corticosteroids within the 28 days prior to and including the first study visit.
* Sinus surgery within 180 days prior to the first study visit

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants for this study will be enrolled into one of two groups. The first group (HEMT Group) will enroll children between 2-8 years of age who have a clinical intent to initiate HEMT, which is defined as ivacaftor or elexacaftor/tezacaftor/ivacaftor based on underlying CFTR mutation status. The second group (non-HEMT Group) will consist of children under the age of 8 without intent to clinically initiate HEMT. Children for both groups will be identified and recruited from cystic fibrosis clinics.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in MRI sinus opacification | Baseline, 1-year, and 2-year follow-up
  Measurement involves calculating percent total sinus opacification (%) using MRI, where sinus contents are differentiated into air and soft tissue/fluid.
Change in olfactory bulb volume | Baseline, 1-year, and 2-year follow-up
  Assessment includes segmenting the olfactory bulb on consecutive coronal slices using MRI, then combining these into a 3-dimensional region. The volume of this region is then calculated in cubic millimeters (mm3).

SECONDARY OUTCOMES:
Change in Pediatric Smell Wheel (PSW) Scores | Baseline, 1-year, and 2-year follow-up
  The PSW test involves children identifying microencapsulated odorants. The score (Range: 0-11) is based on the number of correctly identified smells, with higher scores indicating better olfactory function.
Olfactory Cleft Opacification | Baseline, 1-year, and 2-year follow-up
  Olfactory cleft opacification is quantified by segmenting the olfactory cleft on MRI and applying pixel intensity thresholds to calculate the percentage (%) of opacification.
Change in Brief Questionnaire of Olfactory Disorders (BQOD) Scores | Baseline, 1-year, and 2-year follow-up
  This BQOD is a parent-completed survey for assessing olfactory-specific quality of life (QOL). The survey scores (Range: 0-21) quantify the degree of olfactory QOL impairment, with higher scores indicating greater olfactory QOL impairment.
Change in Sinus and Nasal Quality of Life Survey (SN-5) - Symptom Frequency Domains | Baseline, 1-year, and 2-year follow-up
  SN-5 is a parent-completed survey assessing sinus symptoms and QOL in children. It captures sinus infections, nasal obstruction, allergy symptoms, emotional distress, activity limitations, and overall QOL. For the first five symptom domain questions, scores range 1-7 for each domain, higher scores indicating higher frequency at which symptom affected patient over the past 4 weeks.
Change in Sinus and Nasal Quality of Life Survey (SN-5) - Overall Quality of Life (QOL) Domain | Baseline, 1-year, and 2-year follow-up
  SN-5 is a parent-completed survey assessing sinus symptoms and QOL in children. It captures sinus infections, nasal obstruction, allergy symptoms, emotional distress, activity limitations, and overall QOL. The final question assessing the child's overall QOL as a result of nose or sinus problems is scored on a scale 0-10, with higher scores indicating better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Beswick, MD, Principal Investigator — University of California, Los Angeles
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Vermont, Colchester, Vermont
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
Participant data will be securely stored using REDCap software.

REFERENCES:
- [Derived] Liu CM, Fischer JL, Zemanick ET, Woods JC, Markarian KK, Fain SB, Froh D, Heltshe SL, Hoffman LR, Humphries SM, Kramer EL, Ode KL, Lewis M, Li DA, Mata J, Milla SS, Niedbalski PJ, Sawatzky BD, Sim MS, Sullivan JS, Trout AT, Goss CH, Taylor-Cousar JL, Beswick DM. The impact of highly effective modulator therapy on sinusitis and dysosmia in young children with cystic fibrosis: a prospective study protocol. ERJ Open Res. 2025 Jan 13;11(1):00137-2024. doi: 10.1183/23120541.00137-2024. eCollection 2025 Jan. PMID 39811548